CLINICAL TRIAL: NCT01810783
Title: Interventional, Open-label, Flexible-dose Extension Study of Brexpiprazole in Patients With Schizophrenia
Brief Title: Brexpiprazole in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14644B; 2012-002705-21 (EudraCT Number)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brexpiprazole (Experimental)
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — 1 to 4 mg/day, once daily, tablets, orally. The patients received 2 mg/day brexpiprazole on Day 1. If a patient could not tolerate the 2 mg dose on Day 1, the dose was decreased to 1 mg/day at Day 2. The patients received 1 or 2 mg/day from Days 2 to 7, 1, 2, or 3 mg/day from Days 8 to 14, and 1, 2, 3, or 4 mg/day from Day 15 to completion of the Treatment Period (up-titration).

SUMMARY:
To determine the safety and efficacy of brexpiprazole during long-term treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has completed the lead-in study 14644A.
* The patient is judged to potentially benefit from 52-week treatment with brexpiprazole according to the clinical opinion of the investigator.
* The patient agrees to protocol-defined use of effective contraception.

Exclusion Criteria:

* The patient has been diagnosed with a primary psychiatric disorder other than schizophrenia during Study 14644A.
* The patient has a clinically significant unstable illness diagnosed during Study 14644A.
* The patient, in the opinion of the investigator or according to Columbia-Suicide Severity Rating Scale (C-SSRS), is at significant risk of suicide.
* The patient has an abnormal ECG or other abnormal ECG tests that are, in the investigator's opinion, clinically significant.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (48):
- United States (17):
  - US010, Anaheim, California
  - US020, Cerritos, California
  - US009, Escondido, California
  - US022, Garden Grove, California
  - US018, Long Beach, California
  - US011, San Diego, California
  - US021, Washington D.C., District of Columbia
  - US004, Kissimmee, Florida
  - US015, North Miami, Florida
  - US019, Lake Charles, Louisiana
  - US016, St Louis, Missouri
  - US002, Cedarhurst, New York
  - US005, Charleston, South Carolina
  - US003, Austin, Texas
  - US012, Austin, Texas
  - US001, Dallas, Texas
  - US013, Dallas, Texas
- Estonia (2):
  - EE002, Pärnu
  - EE001, Tallinn
- Poland (3):
  - PL002, Choroszcz
  - PL005, Choroszcz
  - PL004, Gdansk
- Romania (6):
  - RO004, Brasov
  - RO007, Bucharest
  - RO011, Bucharest
  - RO012, Bucharest
  - RO010, Iași
  - RO006, Piteşti
- Russia (7):
  - RU001, Arkhangelsk
  - RU008, Moscow
  - RU015, Rostov-on-Don
  - RU004, Saint Petersburg
  - RU005, Saint Petersburg
  - RU013, Saint Petersburg
  - RU002, Saratov
- Serbia (4):
  - RS001, Belgrade
  - RS003, Belgrade
  - RS002, Kragujevac
  - RS004, Novi Kneževac
- SK001, Liptovský Mikuláš, Slovakia
- Ukraine (8):
  - UA012, Dnipropetrovsk
  - UA004, Geikivka
  - UA007, Hlevakha
  - UA005, Kherson
  - UA008, Kyiv
  - UA009, Lviv
  - UA002, Smila
  - UA003, Vinnytsia

REFERENCES:
- [Derived] Correll CU, He Y, Therrien F, MacKenzie E, Meehan SR, Weiss C, Hefting N, Hobart M. Effects of Brexpiprazole on Functioning in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. J Clin Psychiatry. 2022 Mar 1;83(2):20m13793. doi: 10.4088/JCP.20m13793. PMID 35235720
- [Derived] Marder SR, Meehan SR, Weiss C, Chen D, Hobart M, Hefting N. Effects of Brexpiprazole Across Symptom Domains in Patients With Schizophrenia: Post Hoc Analysis of Short- and Long-Term Studies. Schizophr Bull Open. 2021 May 1;2(1):sgab014. doi: 10.1093/schizbullopen/sgab014. eCollection 2021 Jan. PMID 34901863

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brexpiprazole
Started | 210
Completed | 101
Not Completed | 109
Not completed — Adverse Event | 32
Not completed — Withdrawal by Subject | 22
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 10
Not completed — Protocol Violation | 5
Not completed — Non-compliance with IMP | 4
Not completed — Adminstrative or other reason(s) | 23
Not completed — Enrolled, not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 208
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.89 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 97
Region of Enrollment [Number; unit: participants]
  United States | 50
  Ukraine | 64
  Slovakia | 1
  Serbia | 19
  Russian Federation | 52
  Estonia | 6
  Poland | 9
  Romania | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of treatment-emergent adverse events (TEAEs)
Time Frame: Up to 52 weeks and a safety follow-up by telephone contact or clinic visit after 30 days after the last dose of investigational medicinal product (IMP)
Population: 210 patients were enrolled, only 209 patients were treated with brexpiprazole.TAES is based on these 209 patients
Measure: Number; unit: TEAEs
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 209
TEAEs | 337

ADVERSE EVENTS:
Time Frame: Baseline to end of study
Groups:
- Brexpiprazole: 210 were enrolled, only 209 patients were treated with brexpiprazole
Arm/Group | Brexpiprazole
Serious Adverse Events (participants affected / at risk) | 31/209
Other Adverse Events (participants affected / at risk) | 47/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Brexpiprazole (N=209)
Colitis (Gastrointestinal disorders) | 1
Peritonsillar abscess (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Grand mal convulsion (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/112 — 210 were enrolled, only 209 patients were treated with brexpiprazole, where 112 were women
Aggression (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 2
Schizophrenia (Psychiatric disorders) | 18
Suicidal ideation (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Social stay hospitalisation (Social circumstances) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=209)
Weight increased (Investigations) | 22
Headache (Nervous system disorders) | 18
Insomnia (Psychiatric disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No